CLINICAL TRIAL: NCT00537459
Title: A Randomized, Double-blind, Placebo-controlled, Two-session Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of an 16448 in Healthy Males With Premature Ejaculation.
Brief Title: A Study On Concentrations Of 16448 In Blood And The Safety Of This Compound In Healthy Males With Premature Ejaculation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OTP108172
Record Dates: First submitted 2007-01-25; First posted 2007-10-01 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation (PE) ejaculatory latency time (ELT)
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 16448

SUMMARY:
16448 is being investigated for the treatment of primary premature ejaculation (PE) using a novel mode of action. There are no approved therapies for premature ejaculation, and novel therapies are needed for this syndrome.

16448 has been shown to increase ejaculatory latency in the PCA rat model of premature ejaculation.

A novel instrument, the Sexual Assessment Monitor (SAM), will be used to measure ejaculatory latency time in this study. This device, which measures ELT under standard conditions, has been shown to provide a more reliable measure of ejaculatory latency compared to the use of a stopwatch during sexual intercourse

ELIGIBILITY:
Inclusion criteria:

* Body weight >50kg
* Body Mass Index (BMI): 19-30
* Healthy men with long term (at least 6 months) symptoms of PE
* Erectile Dysfunction - (patients should have EF(Erectile Function) domain of IIEF(International Index of Erectile Function questionnaire >26 or normal)
* No history of reduced sexual desire
* No history of significant psychiatric illness or currently active significant medical illness
* No SSRI's(Selective Serotonin Reuptake Inhibitors) use within the last 4 months
* No history of diabetes, renal or hepatic disease
* No significant injuries to the head or spinal cord i.e. history of head injury, spinal cord injuries, and conditions such as multiple sclerosis.

Exclusion criteria:

* Previous or current use of any PDE-5(Phosphodiesterase type 5) inhibitors for the treatment of Erectile Dysfunction
* Subject receiving treatment in the last 6 months for depression, psychiatric disorders, mood disorders, schizophrenia, substance abuse or anxiety disorders
* Subject is taking tricyclic anti-depressants, selective serotonin reuptake inhibitors (or related drugs), mono-amine oxidase inhibitors or ß-blockers
* Subject has received or is continuing to receive any treatment for PE (e.g. local anaesthetic spray, or intra-cavernosal injection) in the four weeks prior to the study start
* Subject has a history of other clinically significant organic diseases e.g. uncontrolled hypertension, ischemic heart

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
-vital signs, ECGs, clinical laboratory tests, adverse events at 24h -area under plasma drug concentration versus time curve [AUC (0-t),AUC (0-8)], maximum observed plasma concentration (Cmax),time at max concentration(Tmax)& half life (T1/2) | 24h

SECONDARY OUTCOMES:
Measurement of ELT following a single dose of 16448 compared to placebo at approximately 1-2h, post-dose | 1-2h, post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belfast, Ireland